CLINICAL TRIAL: NCT02790606
Title: Prospective, Multi-Center Clinical Study of the Bard® COVERA™ Arteriovenous (AV) Stent Graft in the Treatment of Stenosis at the Graft-Vein Anastomosis of AV Graft Circuits (AVeVA)
Brief Title: Clinical Study of the BARD® COVERA™ Arteriovenous (AV) Stent Graft in AV Graft Patients (AVeVA)
Acronym: AVeVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-15-001
Record Dates: First submitted 2016-05-25; First posted 2016-06-06 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Stenosis; Restenosis
Keywords: ESRD; Stenosis; Restenosis; Hemodialysis; AV Graft
MeSH Terms: conditions — Constriction, Pathologic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: Yes

ARMS (1):
- Covera(TM) Vascular Covered Stent (Experimental): Placement of the Covera Vascular Covered Stent following percutaneous transluminal angioplasty (PTA)
  Interventions: Device: Covera(TM) Vascular Covered Stent

INTERVENTIONS:
Device: Covera(TM) Vascular Covered Stent — Treatment of stenoses with primary percutaneous transluminal angioplasty (PTA) and placement of the Covera Vascular Covered Stent.

SUMMARY:
The objective of this study is to assess the safety and effectiveness of the COVERA™ Vascular Covered Stent for the treatment of stenotic lesions in the upper extremity venous outflow of the Arteriovenous (AV) access circuit.

DETAILED DESCRIPTION:
This study will compare the use of the COVERA™ Vascular Covered Stent (following percutaneous transluminal angioplasty (PTA)) to safety and effectiveness performance goals (PGs) for the treatment of stenotic lesions in the upper extremity venous outflow of the arteriovenous (AV) access circuit of subjects dialyzing with an AV graft.

ELIGIBILITY:
Clinical Inclusion Criteria:

* Subject must voluntarily sign and date the Informed Consent Form (ICF) prior to collection of study data or performance of study procedures.
* Subject must be either a male or non-pregnant female ≥ 21 years of age with an expected lifespan sufficient to allow for completion of all study procedures.
* Subject must be willing to comply with the protocol requirements, including clinical and telephone follow-up.
* Subject must have a synthetic AV access graft located in an arm that has been implanted for ≥ 30 days and must have undergone at least one successful dialysis session prior to the index procedure.

Angiographic Inclusion Criteria

* Subject must have angiographic evidence of a stenosis ≥ 50% (by visual estimation) located at the graft-vein anastomosis of the subject's synthetic AV access graft and present with clinical evidence of graft dysfunction at the synthetic AV graft-vein anastomosis.
* The target lesion must be ≤ 9cm in length. Note: multiple stenoses may exist within the target lesion.
* The reference vessel diameter of the adjacent non-stenotic vessel must be between 5.0 and 9.0mm.

Clinical Exclusion Criteria:

* The subject is dialyzing with an AV fistula.
* The hemodialysis access is located in the lower extremity.
* The subject has an infected AV access graft or uncontrolled systemic infection.
* The subject has a known uncontrolled blood coagulation/bleeding disorder.
* The subject has a known allergy or hypersensitivity to contrast media which cannot be adequately pre-medicated.
* The subject has a known hypersensitivity to nickel-titanium (Nitinol) or tantalum.
* The subject has another medical condition, which, in the opinion of the Investigator, may cause him/her to be non-compliant with the protocol, confound the data interpretation, or is associated with a life expectancy insufficient to allow for the completion of study procedures and follow-up.
* The subject is currently participating in an investigational drug or another device study that has not completed the study treatment or that clinically interferes with the study endpoints. Note: Studies requiring extended follow-up visits for products that were investigational, but have since become commercially available, are not considered investigational studies.

Angiographic Exclusion Criteria:

* Additional stenotic lesions (≥ 50%) in the venous outflow that are > 3cm from the edge of the target lesion and are not successfully treated (defined as < 30% residual stenosis) prior to treating the target lesion.
* An aneurysm or pseudoaneurysm is present within the target lesion.
* The location of the target lesion would require the COVERA™ Vascular Covered Stent be deployed across the elbow joint.
* The target lesion is located within a stent or stent graft.
* The location of the target lesion would require that the COVERA™ Vascular Covered Stent be placed in the central veins (subclavian, brachiocephalic, Superior Vena Cava (SVC)) or under the clavicle at the thoracic outlet.
* There is incomplete expansion of an appropriately-sized angioplasty balloon to its expected profile, in the operator's judgment, during primary angioplasty at the target lesion prior to implantation of the study device.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Dolmatch, M.D., Principal Investigator — The Palo Alto Medical Foundation
Locations (16):
- United States (16):
  - Arizona Kidney Disease and Hypertension Center, Phoenix, Arizona
  - Southwest Vascular Center, Tempe, Arizona
  - Arizona Kidney Disease and Hypertension Center Medical Research Services, LLC, Tucson, Arizona
  - St. Joseph Hospital, Orange, California
  - Capital Nephrology Access Center, Sacramento, California
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Ocala Kidney Group, Ocala, Florida
  - Chicago Access Care, Chicago, Illinois
  - Renal and Transplant Associates of New England, P.C., West Springfield, Massachusetts
  - The Cardiovascular Care Group, Westfield, New Jersey
  - Surgical Specialists of Charlotte, Charlotte, North Carolina
  - NC Heart and Vascular Research, Raleigh, North Carolina
  - NC Nephrology, Raleigh, North Carolina
  - Providence Access Care, Providence, Rhode Island
  - Tarrant Vascular Clinic, Fort Worth, Texas
  - Clinical Advancement Center, PLLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 14 active sites in the US. Of 181 consented subjects,110 were treated with device and 71 were considered screen failures. No site treated more than 20% of the total number of subjects.The first subject was treated Aug, 3, 2016 and the last one Feb. 27, 2017. The last 24-month follow-up contact occurred Mar. 16, 2019.
Groups:
- Covera(TM) Vascular Covered Stent: Vascular Covered Stent for the treatment of stenotic lesions at the graft-vein anastomosis of hemodialysis patients dialyzing with an AV graft.
Period: Overall Study
Arm/Group | Covera(TM) Vascular Covered Stent
Started | 110
Completed (The Milestone is all participants who completed the study (24-month Follow-Up).) | 75
Not Completed | 35
Not completed — Death | 27
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Eight (8) of the 110 enrolled participants have not completed the trial and may therefore not be accounted for in the different follow-up periods, resulting in a discrepancy between the N and n for each period.
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 110
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 52
  ≥ 65 and < 75 years | 31
  ≥ 75 years | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60
  Male | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 86
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 44
  White | 60
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 110
Hemodialysis - Baseline [Mean (Standard Deviation); unit: Months on hemodialysis] — The average number of months on dialysis prior to the index procedure.
  Months on hemodialysis | 19.7 (19.95)
AV Access Circuit Description/ Target Limb [Count of Participants; unit: Participants]
  Left Arm | 88
  Right Arm | 22
AV Access Circuit Description: Graft Location [Count of Participants; unit: Participants]
  Forearm | 2
  Upper Arm | 108
AV Access Circuit Description: Arterial Anastomosis [Count of Participants; unit: Participants]
  Axillary | 14
  Brachial | 94
  Radial | 1
  Ulnar | 1
AV Access Circuit Description: Venous Anastomosis [Count of Participants; unit: Participants]
  Axillary | 54
  Basilic | 44
  Brachial | 9
  Cephalic | 2
  Median Cubital | 1
AV Access Circuit Description: Graft Configuration [Count of Participants; unit: Participants]
  Loop | 33
  Straight | 77
AV Access Circuit Description: Graft Material [Count of Participants; unit: Participants]
  Bovine | 10
  ePTFE | 85
  Other | 4
  Unknown | 11
AV Access Circuit Description: Graft Tapered [Count of Participants; unit: Participants]
  Yes | 32
  No | 78
AV Access Circuit Description: Graft Diameter (mm) [Mean (Standard Deviation); unit: mm] — Population: For three (3) subjects the diameter of the graft at the time of initial access creation on was unknown.
  mm
    number analyzed (Participants) | 107
    (all) | 6.6 (0.77)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From AV Access Circuit Localized or Systemic Serious Adverse Events
Description: Safety is defined as freedom from any adverse event(s) (AEs), localized or systemic, that reasonably suggests the involvement of the AV access circuit (not including stenosis or thrombosis) that require or result in any of the following alone or in combination: additional interventions (including surgery); in-patient hospitalization or prolongation of an existing hospitalization; or death.
Time Frame: 30 days post index procedure
Population: Number of Participants Free from Primary Safety Events (All Treated Subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 110
Participants | 106
Statistical Analysis 1: Comparison: Covera(TM) Vascular Covered Stent; The primary safety endpoint is evaluated against a PG of 88%, which was derived from safety event rates of PTA in published literature. Hypothesis: The safety rate in subjects treated with the COVERA™ Vascular Covered Stent (following PTA) at 30 days post-index procedure is greater than that of the PG of 88%. 109 treated subjects [104 evaluable] will give 99% power with one-sided type I error = 0.05; Test type: Superiority; p = 0.0021, Exact binomial test

2. Primary Outcome: Effectiveness Endpoint: Number of Participants With Target Lesion Primary Patency
Description: Target Lesion Primary Patency (TLPP) is defined as the interval following the index intervention until the next clinically driven reintervention at the original treatment site or until the extremity is abandoned for permanent access.
  Primary patency ends when any of the following occurs: a) clinically driven reintervention in the treatment area; b) thrombotic occlusion within the treatment area; c) surgical intervention that excludes the original treatment area from the AV circuit, and/or d) abandonment of the AV access graft due to inability to treat the original treatment area.
  The primary effectiveness endpoint is evaluated against a performance goal (PG) of 40%.
Time Frame: 6 months post index procedure
Population: Number of participants with Target Lesion Primary Patency.
  In total, nine (9) subjects were excluded from the denominator (110) due to discontinuation or abandonment of their index AV access circuit for non effectiveness reasons prior to Day 150 of their follow-up. Therefore, the Overall Number of Participants analyzed is 101 for this measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 101
Participants | 71
Statistical Analysis 1: Comparison: Covera(TM) Vascular Covered Stent; The primary effectiveness endpoint is evaluated against a PG of 40%, which was derived from clinical literature as well as other pivotal and post-market studies of stent grafts at the graft-vein anastomosis of AV access patients dialyzing with an AV graft. 89% estimated power for primary endpoint. Hypothesis: The proportion of subjects treated with the COVERA™ Vascular Covered Stent (following PTA) with respect to TLPP through 6 months post-index procedure is greater than that of the PG of 40%; Test type: Superiority; p < 0.0001, Exact binomial test — The p-value is compared to the PG (40%) and computed using the exact binomial test

3. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Target Lesion Primary Patency (TLPP)
Description: TLPP is defined as the interval following the index intervention until the next clinically driven reintervention at the original treatment site or until the extremity is abandoned for permanent access.
  Primary patency ends when any of the following occurs: a) clinically driven reintervention in the treatment area; b) thrombotic occlusion within the treatment area; c) surgical intervention that excludes the original treatment area from the AV circuit, and/or d) abandonment of the AV access graft due to inability to treat the original treatment area.
  The 1, 3, 6, 12, 18 and 24 months final results are reported below.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: Number of Participants with Target Lesion Primary Patency.
  Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 30 days, 3 months and 6 months follow-up or did not meet endpoint inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 109
Participants
  TLPP at 30-days Follow-Up | 100
  TLPP at 90-days Follow-up: number analyzed (Participants) | 105
  TLPP at 90-days Follow-up | 91
  TLPP at 6-month Follow-Up: number analyzed (Participants) | 101
  TLPP at 6-month Follow-Up | 71
  TLPP at 12-month Follow-Up: number analyzed (Participants) | 91
  TLPP at 12-month Follow-Up | 46
  TLPP at 18-month Follow-Up: number analyzed (Participants) | 86
  TLPP at 18-month Follow-Up | 33
  TLPP at 24-month Follow-Up: number analyzed (Participants) | 83
  TLPP at 24-month Follow-Up | 25

4. Secondary Outcome: Endpoint With Hypothesis Testing: Number of Participants With Access Circuit Primary Patency (ACPP)
Description: ACPP is defined as the interval following the index intervention until the next access thrombosis or repeated intervention.
  ACPP ends with a reintervention anywhere within the access circuit. Vessel rupture caused by PTA is not an ACPP failure unless achieving hemostasis also causes thrombosis.
  The 1, 3, 6, 12, 18 and 24 months final results are reported below.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: Number of Participants with Access Circuit Primary Patency (ACPP).
  Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 30 days, 3 months and 6 months follow-up or did not meet endpoint inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 109
Participants
  ACPP at 30-days Follow-Up | 96
  ACPP at 90-days Follow-Up: number analyzed (Participants) | 106
  ACPP at 90-days Follow-Up | 72
  ACPP at 6-months Follow-Up: number analyzed (Participants) | 102
  ACPP at 6-months Follow-Up | 40
  ACPP at 12-months Follow-Up: number analyzed (Participants) | 97
  ACPP at 12-months Follow-Up | 14
  ACPP at 18-months Follow-Up: number analyzed (Participants) | 94
  ACPP at 18-months Follow-Up | 7
  ACPP at 24-months Follow-Up: number analyzed (Participants) | 94
  ACPP at 24-months Follow-Up | 4

5. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Device and Procedure Related AEs Involving the AV Access Circuit
Description: Number of Participants with device and procedure related Adverse Events involving the AV access circuit.
  The access circuit is the area from the arterial inflow to the SVC-right atrial junction.
  The 1, 3, 6, 12, 18 and 24 months final results are reported below.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure,
Population: Number of Participants Free from Device/Procedure-Related Adverse Events.
  Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 30 days, 3 months and 6 months follow-up or did not meet endpoint inclusion criteria.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 110
Participants
  30-days Follow-Up | 105
  90-days Follow-Up: number analyzed (Participants) | 108
  90-days Follow-Up | 99
  6-months Follow-Up: number analyzed (Participants) | 105
  6-months Follow-Up | 96
  12-months Follow-Up: number analyzed (Participants) | 96
  12-months Follow-Up | 85
  18-months Follow-Up: number analyzed (Participants) | 88
  18-months Follow-Up | 77
  24-months Follow-Up: number analyzed (Participants) | 80
  24-months Follow-Up | 69

6. Secondary Outcome: Endpoint Without Hypothesis Testing: Total Number of Arteriovenous (AV) Access Circuit Reinterventions
Description: Total Number of AV Access Circuit Reinterventions defined as the number of reinterventions to the AV access circuit until access abandonment or through study completion.
  The 1, 3, 6, 12, 18 and 24 months final results are reported below.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure.
Population: Total number of AV Access Circuit Reinterventions by Follow-Up Period. The number for a specific period may be higher than the number of subjects with at least one AV access reintervention in that period. Number of participants (n) varies from overall enrollment (N) due to discontinued participation or not meeting endpoint inclusion criteria.
Measure: Number; unit: AV Access Reinterventions
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 108
AV Access Reinterventions
  AV Access Circuit Reinterventions at 30 days | 16
  AV Access Circuit Reinterventions at 90 days: number analyzed (Participants) | 105
  AV Access Circuit Reinterventions at 90 days | 51
  AV Access Circuit Reinterventions at 6-months: number analyzed (Participants) | 101
  AV Access Circuit Reinterventions at 6-months | 111
  AV Access Circuit Reinterventions at 12-months: number analyzed (Participants) | 96
  AV Access Circuit Reinterventions at 12-months | 222
  AV Access Circuit Reinterventions at 18-months: number analyzed (Participants) | 93
  AV Access Circuit Reinterventions at 18-months | 284
  AV Access Circuit Reinterventions at 24-months: number analyzed (Participants) | 93
  AV Access Circuit Reinterventions at 24-months | 333

7. Secondary Outcome: Endpoint Without Hypothesis Testing: Total Number of Target Lesion Reinterventions
Description: Total Number of Target Lesion Reinterventions defined as the number of reinterventions to maintain target lesion patency.
  The 1, 3, 6, 12, 18 and 24 months final results are reported below.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: The (n) in each follow-up periods vary from overall enrollment (N) as some subjects discontinued participation before each follow-up or did not meet endpoint inclusion criteria.
  The total number of Reinterventions by Follow-Up Period was analyzed as opposed to the number of subjects with at least one AV Target Lesion Reintervention.
Measure: Number; unit: Target Lesion Reinterventions
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 108
Target Lesion Reinterventions
  Target Lesion Reintervention at 30 days Follow-Up | 10
  Target Lesion Reintervention at 90 days Follow-Up: number analyzed (Participants) | 104
  Target Lesion Reintervention at 90 days Follow-Up | 18
  Target Lesion Reintervention at 6 months Follow-Up: number analyzed (Participants) | 100
  Target Lesion Reintervention at 6 months Follow-Up | 44
  Target Lesion Reintervention at 12 month Follow-Up: number analyzed (Participants) | 89
  Target Lesion Reintervention at 12 month Follow-Up | 81
  Target Lesion Reintervention at 18 month Follow-Up: number analyzed (Participants) | 80
  Target Lesion Reintervention at 18 month Follow-Up | 100
  Target Lesion Reintervention at 24 month Follow-Up: number analyzed (Participants) | 75
  Target Lesion Reintervention at 24 month Follow-Up | 116

8. Secondary Outcome: Endpoint Without Hypothesis Testing: Index of Patency Function (IPF)
Description: IPF is defined as the time from the index study procedure to study completion or access abandonment divided by the number of visits for a reintervention performed on the AV access circuit in order to maintain vascular access for hemodialysis.
  The 1, 3, 6, 12, 18 and 24 months final results are reported below.
  The IPF is representative of the number of days between interventions to maintain access circuit patency. The minimum and maximum ranges for the Index of Patency Function are as follows: 1 month (6.3 - 30.0); 3 months (6.3 - 90.0); 6 months (6.3 - 180.0); 12 months (6.3 - 365.0); 18 months (6.3 - 545.0); and 24 months (6.3 - 730.0). Higher values represent a better outcome, that is, more time elapsed between the Index study procedure and reinterventions.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: Number of participants (n) in each follow-up periods varies from overall enrollment (N) as some subjects discontinued participation before the 30 days, 3 months and 6 months follow-up or did not meet endpoint inclusion criteria.
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 108
Index
  Index of Patency Function at 30 days Follow-Up | 28.10 (5.446)
  Index of Patency Function at 90 days Follow-Up: number analyzed (Participants) | 105
  Index of Patency Function at 90 days Follow-Up | 72.24 (26.01)
  Index of Patency Function at 6 months Follow-Up: number analyzed (Participants) | 101
  Index of Patency Function at 6 months Follow-Up | 110.3 (57.71)
  Index of Patency Function at 12 months Follow-Up: number analyzed (Participants) | 96
  Index of Patency Function at 12 months Follow-Up | 144.3 (102.6)
  Index of Patency Function at 18 months Follow-Up: number analyzed (Participants) | 93
  Index of Patency Function at 18 months Follow-Up | 163.1 (131.6)
  Index of Patency Function at 24 months Follow-Up: number analyzed (Participants) | 93
  Index of Patency Function at 24 months Follow-Up | 177.9 (153.2)

9. Secondary Outcome: Endpoint Without Hypothesis Testing: Index of Patency Function - Target Lesion (IPF-T)
Description: IPF-T (Index of Patency Function - Target Lesion) is defined as the time from the index study procedure to study completion or complete access abandonment divided by the number of visits for a reintervention performed at the target lesion in order to maintain vascular access for hemodialysis.
  The 1, 3, 6, 12, 18 and 24 months final results are reported below.
  The IPF for target lesion patency is representative of the approximate (mean) number of days between interventions to maintain target lesion patency. The minimum and maximum ranges for the Index of Patency Function are as follows: 1 month (6.3 - 30.0); 3 months (6.3 - 90.0); 6 months (6.3 - 180.0); 12 months (6.3 - 365.0); 18 months (6.3 - 545.0); and 24 months (6.3 - 730.0). Higher values represent a better outcome, that is, more time elapsed between the Index study procedure and reinterventions.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 108
Index
  IPTF-T at 30 days Follow-Up | 28.75 (4.475)
  IPTF-T at 90 days Follow-Up: number analyzed (Participants) | 104
  IPTF-T at 90 days Follow-Up | 83.27 (18.48)
  IPTF-T at 6 months Follow-Up: number analyzed (Participants) | 100
  IPTF-T at 6 months Follow-Up | 146.3 (52.30)
  IPTF-T at 12 months Follow-Up: number analyzed (Participants) | 89
  IPTF-T at 12 months Follow-Up | 253.2 (127.3)
  IPTF-T at 18 months Follow-Up: number analyzed (Participants) | 80
  IPTF-T at 18 months Follow-Up | 325.7 (197.3)
  IPTF-T at 24 months Follow-Up: number analyzed (Participants) | 75
  IPTF-T at 24 months Follow-Up | 380.3 (270.7)

10. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Post-intervention Secondary Patency
Description: Secondary Patency is defined as the interval after the index intervention until the access is abandoned. Multiple repetitive treatments can be included in post-intervention secondary patency.
  The 1, 3, 6, 12, 18 and 24 months final results are reported below.
Time Frame: 1, 3, 6, 12, 18 and 24 months post index procedure
Population: Post-Intervention Secondary Patency by Follow-Up Period (All Treated Subjects).
  (n) varies in relation to the number of failures (access abandonment) recorded at 30 days, 90 days and 6 months. Accordingly, the (n) for each period may be different from the overall (N) reported in the Participant Flow section.
Measure: Count of Participants; unit: Participants
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 109
Participants
  Participants with Secondary Patency at 30 days | 107
  Participants with Secondary Patency at 90 days: number analyzed (Participants) | 105
  Participants with Secondary Patency at 90 days | 101
  Participants with Secondary Patency at 6 months: number analyzed (Participants) | 101
  Participants with Secondary Patency at 6 months | 93
  Participants with Secondary Patency at 12 months: number analyzed (Participants) | 89
  Participants with Secondary Patency at 12 months | 76
  Participants with Secondary Patency at 18 months: number analyzed (Participants) | 80
  Participants with Secondary Patency at 18 months | 64
  Participants with Secondary Patency at 24 months: number analyzed (Participants) | 72
  Participants with Secondary Patency at 24 months | 53

11. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Technical Success (for Stent Graft Placement)
Description: Technical Success is defined as successful deployment, based on the operator's opinion, of the implant to the intended location assessed at the time of the index procedure.
Time Frame: At time of index procedure
Population: Number of Participants with Acute Technical Success (All Treated Subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 110
Participants | 110

12. Secondary Outcome: Endpoint Without Hypothesis Testing: Number of Participants With Procedure Success
Description: Procedure Success is defined as anatomic success and resolution of the pre-procedural clinical indicator(s) (clinical success) of a hemodynamically significant stenosis.
Time Frame: At time of index procedure
Population: Procedure Success (All Treated Subjects)
Measure: Count of Participants; unit: Participants
Arm/Group | Covera(TM) Vascular Covered Stent
Number analyzed (Participants) | 110
Participants | 110

ADVERSE EVENTS:
Time Frame: Adverse events experienced by subjects were collected during a 24-month follow-up period (from the index procedure through the final follow-up contact, or early termination).
Description: Adverse events collection was limited to localized or systemic clinical manifestations that reasonably suggests involvement of the AV access circuit (related to graft to the SVC-right atrial junction).
  Systematic assessment was achieved through scheduled phone calls (or in-office visits) at 30 days, 90 days, 6 months, 12 months, 18 months and 24 months post procedure.
Arm/Group | Covera(TM) Vascular Covered Stent
All-Cause Mortality (participants affected / at risk) | 27/110
Serious Adverse Events (participants affected / at risk) | 41/110
Other Adverse Events (participants affected / at risk) | 53/110
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Covera(TM) Vascular Covered Stent (N=110)
Arteriovenous Graft Site Infection (Infections and infestations) | 7
Vascular Graft Complication (Injury, poisoning and procedural complications) | 22
Arteriovenous Fistula (Vascular disorders) | 1
Steal Syndrome (Vascular disorders) | 3
Vascular Rupture (Vascular disorders) | 1
Vasospasm (Vascular disorders) | 1
Infusion Site Extravasation (General disorders) | 4
Stent Malfunction (General disorders) | 1
Infected Skin Ulcer (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Arteriovenous Graft Aneurysm (Injury, poisoning and procedural complications) | 4
Arteriovenous Graft Site Haemorrhage (Injury, poisoning and procedural complications) | 2
Seroma (Injury, poisoning and procedural complications) | 1
Skin Wound (Injury, poisoning and procedural complications) | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 5
Vascular Dissection (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Covera(TM) Vascular Covered Stent (N=110)
Local Swelling (General disorders) | 1
Arteriovenous Graft Site Infection (Infections and infestations) | 7
Arteriovenous Graft Site Haemorrhage (Injury, poisoning and procedural complications) | 3
Vascular Graft Complication (Injury, poisoning and procedural complications) | 30
Paraesthesia (Nervous system disorders) | 1
Arteriovenous Fistula (Vascular disorders) | 1
Steal Syndrome (Vascular disorders) | 5
Vascular Rupture (Vascular disorders) | 1
Vasospasm (Vascular disorders) | 1
Infusion Site Extravasation (General disorders) | 4
Stent Malfunction (General disorders) | 1
Infected Skin Ulcer (Infections and infestations) | 1
Wound Infection (Infections and infestations) | 1
Arteriovenous Graft Aneurysm (Injury, poisoning and procedural complications) | 4
Arteriovenous Graft Site Haematoma (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Skin Wound (Injury, poisoning and procedural complications) | 1
Vascular Pseudoaneurysm (Injury, poisoning and procedural complications) | 6
Vascular Dissection (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to PI publication of site results, sponsor requires publication of multi-centers results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-03): https://cdn.clinicaltrials.gov/large-docs/06/NCT02790606/Prot_SAP_000.pdf